CLINICAL TRIAL: NCT03862027
Title: Evaluating Safety of Transpulmonary Pressure Guided PEEP Management in Neurocritical Care Patients
Brief Title: Safety of Optimal PEEP in NSICU Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to enroll/recruit
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-2064
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2020-09

CONDITIONS: Respiratory Failure; Intracranial Hypertension
MeSH Terms: conditions — Respiratory Insufficiency; Intracranial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Esophageal Balloon catheter (Experimental): All patients will have an esophageal balloon catheter inserted into their nare while upright (head of bed > 30 degrees) to a depth slightly more than the estimated distance from the lower sternum to the back of the ear (typically around 60 cm). Gastric positioning will be confirmed with abdominal compression testing and the catheter then retracted 10 - 20 cm into the lower esophagus. Placement will be confirmed with the presence of cardiac oscillations on the esophageal probe. The probe will then be secured to the patient's nasal opening using tape.
  Interventions: Device: Esophageal Balloon catheter

INTERVENTIONS:
Device: Esophageal Balloon catheter — Pressures [Esophageal Pressure (Pes), Airway Pressure (Paw), and Transpulmonary Pressure (Ptp)] are measured directly through the ventilator. The waveforms of Paw, Pes, and Ptp will be visualized on the ventilator. Ptp is obtained from Paw - Pes. All patients will have baseline measurements recorded of ICP, CPP, and MAP.
  PEEP will be increased on the ventilator to achieve a Ptp between 0 and +2 cm H2O ("Optimal PEEP").
  Measurements of Intracranial pressure (ICP), cerebral perfusion pressure (CPP), and mean arterial pressure (MAP) will be repeated 5 minutes after the change in PEEP.

SUMMARY:
The investigators aim to demonstrate that use of transpulmonary pressure to guide PEEP management is safe in patients with possible elevations of intracranial pressure.

DETAILED DESCRIPTION:
Purpose: To establish safety of titrating PEEP based on transpulmonary pressure as measured by an esophageal balloon in mechanically ventilated neurosurgical patients.

Participants: Adult patients admitted to the Neuro ICU at UNC Hospital and requiring mechanical ventilation who have an intracranial pressure monitoring device in place.

Procedures (methods): All enrolled patients will have esophageal balloons placed with measurement of transpulmonary pressures. All patients will have baseline measurements recorded of intracranial pressure, cerebral perfusion pressure, and cerebral autoregulation. PEEP will then be titrated based on transpulmonary pressure measurements with recording of physiological measurements over the next hour. At the conclusion of the hour, all patients will be returned to their prior ventilator settings.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >/= 18) admitted to the Neuro ICU of UNC Hospital requiring mechanical ventilation and with ICP monitoring in place.

Exclusion Criteria:

1. Pneumothorax or pneumomediastinum
2. Life expectancy < 24 hours or expected to require mechanical ventilation for < 24 hours
3. Condition that precludes placement of an esophageal balloon [esophageal or nasopharyngeal pathology preventing insertion of the esophageal balloon catheter (esophageal ulcerations, tumors, diverticulitis, bleeding varices or in patients with sinusitis, epistaxis or recent nasopharyngeal surgery), severe thrombocytopenia (platelet count < 30) or coagulopathy (INR > 3 or on oral anticoagulants).
4. Pre-enrollment ICP > 20 mm Hg
5. Pre-enrollment CPP < 60 mm Hg
6. Planned change in the external ventricular drain set point during the pre-intervention, intervention or post-intervention periods
7. Incarceration
8. Variation in ICP of > 2 cm H2O in the hour prior to intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Carson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Esophageal Balloon Catheter: All patients will have an esophageal balloon catheter inserted into their nare while upright (head of bed > 30 degrees) to a depth slightly more than the estimated distance from the lower sternum to the back of the ear (typically around 60 cm). Gastric positioning will be confirmed with abdominal compression testing and the catheter then retracted 10 - 20 cm into the lower esophagus. Placement will be confirmed with the presence of cardiac oscillations on the esophageal probe. The probe will then be secured to the patient's nasal opening using tape.
  Esophageal Balloon catheter: Pressures [Esophageal Pressure (Pes), Airway Pressure (Paw), and Transpulmonary Pressure (Ptp)] are measured directly through the ventilator. The waveforms of Paw, Pes, and Ptp will be visualized on the ventilator. Ptp is obtained from Paw - Pes. All patients will have baseline measurements recorded of ICP, CPP, and MAP.
  PEEP will be increased on the ventilator to achieve a Ptp between 0 and +2 cm H2O ("Optimal PEEP").
  Measurements of Intracranial pressure (ICP), cerebral perfusion pressure (CPP), and mean arterial pressure (MAP) will be repeated 5 minutes after the change in PEEP.
Period: Overall Study
Arm/Group | Esophageal Balloon Catheter
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Esophageal Balloon Catheter
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in ICP Value
Description: The Intracranial pressure (ICP) value after intervention will be considered equivalent to the ICP before intervention if the 95% upper bound of the change is lower than the non-inferiority margin of 4 mm Hg.
Time Frame: Within 5 minutes of catheter placement
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Esophageal Balloon Catheter
Number analyzed (Participants) | 1
mm Hg | 0 (NA) — Standard Deviation not derived because n=1

2. Secondary Outcome: Change in Cerebral Perfusion Pressure (CPP)
Description: Cerebral perfusion pressure is equal to the mean arterial pressure (MAP) minus the intracranial pressure (ICP). The initial CPP is calculated by measuring CPP immediately before changing ventilator settings. The post-intervention CPP is measured 5 minutes after ventilator setting change is made. The difference between the initial CPP and the post-intervention CPP reflects the change in CPP.
Time Frame: Immediately before and 5 minutes after ventilator setting change
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Esophageal Balloon Catheter
Number analyzed (Participants) | 1
mm Hg | 1 (NA) — Standard Deviation not derived because n=1

3. Secondary Outcome: Change in Mean Arterial Pressure
Description: Mean Arterial Pressure (MAP) is the average arterial pressure in one cardiac cycle measured through an arterial line.
Time Frame: Immediately before and 5 minutes after ventilator setting change
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Esophageal Balloon Catheter
Number analyzed (Participants) | 1
mm Hg | 1 (NA) — Standard Deviation not derived because n=1

ADVERSE EVENTS:
Time Frame: From the time of procedure through 24 hours afterwards.
Arm/Group | Esophageal Balloon Catheter
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT03862027/Prot_SAP_000.pdf